CLINICAL TRIAL: NCT03211962
Title: Can Urinary Concentrations of TIMP2 and IGFBP7 be Used to Predict Early Acute Renal Failure Following Cardiac Arrest?
Acronym: ACR-CHECK
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2015-09
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Renal Failure; Heart Failure
MeSH Terms: conditions — Renal Insufficiency; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analysis of urinary levels of TIMP2 and IGFBP7 within 6 hours after cardiac circulatory arrest — Analysis of urinary levels of TIMP2 and IGFBP7 within 6 hours after cardiac circulatory arrest

SUMMARY:
Transient renal insufficiency is frequently observed in the course of cardiovascular arrest. Although elevation of creatinine is reversible in a large majority of cases, severe renal insufficiency is sometimes observed and is associated with a dark prognosis. Any intervention that may limit the worsening of renal function may have an impact on patient mortality. There is currently no validated pharmacological treatment to limit the progression of ARI or to accelerate its recovery. A major challenge then concerns the detection of the reversible character of renal damage.

Renal biomarkers have been little studied in the prediction of severe ARI and mortality after cardiac arrest. The combination of TIMP2 (tissue inhibitor of metalloproteinase) and insulin-like growth factor binding protein (IGFBP7) in urine showed good diagnostic performance in the early detection of the risk of developing acute renal failure within 12 hours. Measured in the urine, the excretion of these two markers specifically reflects renal tubular lesions. Moreover, their rate seems to be strongly correlated with the severity of the tubular lesions.

Thus, it can be reasonably assumed that their very early dosing in post-cardiac arrest could detect the presence and severity of renal tubular lesions. A threshold to be defined would discriminate patients at risk of developing an ARI within 48 hours post ACR and to distinguish between severe transient and severe persistent lesions beyond 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Cardio-circulatory arrest within 6 hours
* Person affiliated to a social security scheme

Exclusion Criteria:

* Acute renal failure requiring urgent ERA in the opinion of the resuscitator Anuria
* Chronic renal insufficiency stage 4-5 with a glomerular filtration rate estimated at less than 30 ml / min.
* Rapidly progressive renal disease (glomerulonephritis, HUS, obstruction ...) Renal Insufficiency
* Probable glomerular involvement (nephritic syndrome, nephrotic syndrome, chronic glomerulonephritis)
* Pregnant or nursing women
* Patient under tutelage or curatorship or deprived of public right.
* Transplantation
* Subject involved in another search including an exclusion period still in progress at pre-inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to resuscitation in the aftermath of cardiac arrest with renal failure
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Analysis of the predictive value of the urinary concentration of TIMP2-IGFBP7 | Analysis of the predictive value of the urinary concentration of TIMP2-IGFBP7 in the development of acute renal insufficiency defined by the KDIGO 3 stage within 48 hours after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France